CLINICAL TRIAL: NCT06228391
Title: Examining the Efficacy and Safety of Subanesthetic Ketamine on Depression and Post-traumatic Stress Among Veterans With Mild and Moderate Traumatic Brain Injury
Brief Title: Ketamine Treatment for PTSD and MDD in TBI
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Paulo Shiroma, Psychiatrist, Minneapolis Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1770474-4
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: PTSD, Post Traumatic Stress Disorder; Major Depressive Disorder; Traumatic Brain Injury
Keywords: Veteran; Ketamine; PTSD; Depression; TBI
MeSH Terms: conditions — Combat Disorders; Depressive Disorder, Major; Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic; Depression | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ketamine (Experimental): Twice a week ketamine IV 0.5 mg/kg
  Interventions: Drug: IV ketamine
- Midazolam (Active Comparator): Twice a week midazolam IV 0.045 mg/kg
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: IV ketamine — Subjects will receive a single infusion of racemic ketamine at 0.5mg/kg for 40 minutes twice a week for 3 weeks.
  Arms: Ketamine
Drug: Midazolam — Subjects will receive a single infusion of midazolam at 0.045mg/kg for 40 minutes twice a week for 3 weeks.
  Arms: Midazolam

SUMMARY:
The goal of this clinical trial is to examine the use of sedative ketamine to treat depression and post-traumatic stress disorder (PTSD) in Veterans with mild to moderate traumatic brain injury (TBI). The main questions it aims to answer are:

* Efficacy of ketamine to reduce symptoms of depression and/or PTSD
* Safety of ketamine to treat depression and/or PTSD in TBI Participants will be randomly assigned to receive either ketamine or midazolam (active placebo) twice a week for 3 weeks. During participation, subjects will be interviewed, have lab tests, and complete rating scales, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Willingness/able to sign informed consent.
* Able to read and write in English.
* Male or female Veterans aged 18-55 years old.
* Remote history of TBI mild-moderate that is ≥12 weeks post-injury (chronic period) that met at minimum the 2021 VA/DoD Clinical Practice Guideline for the Management and Rehabilitation of Post-Acute Mild Traumatic Brain Injury (i.e., new onset or worsening of at least one of the following clinical signs immediately following the event: loss or decreased of consciousness, period of posttraumatic amnesia, period of being dazed and confused, and neurologic deficits).
* Lifetime history of treatment resistance to at least one adequate trial of an antidepressant as determined by the Massachusetts General Hospital Antidepressant Treatment History Questionnaire (MGH-ATRQ).
* FDA-approved antidepressant, trazodone, atypical neuroleptic, prazosin, or clonidine with stable treatment, as determined by the study clinician, for at least 4 weeks prior to randomization. Following randomization, changes to doses may be allowable at the investigator's discretion

Exclusion Criteria:

* Ketamine treatment within the last 6 months

  * Lifetime history of psychosis-related disorder, current episode of mania/hypomania/mixed assessed by the Mini-International Neuropsychiatric Interview (MINI 7.0 for DSM-5).
  * History of penetrating head wounds or severe traumatic brain injury (Glasgow Coma Scale <9; loss of consciousness >24hr; post-traumatic amnesia>7 days).
  * Severe substance and/or alcohol use disorder (DSM-5-TR) within six months of initial assessment; presence of illicit drugs (except cannabis) by positive urine toxicology at screening.
  * Intellectual disability or pervasive developmental disorder; dementia of any type.
  * Any disorder that, based on the Principal Investigator's judgement, would increase risk (e.g., unstable cardiac conditions) or protocol adherence (e.g., severe personality disorder).
  * For women: pregnancy (confirmed by lab test), initiation of female hormonal treatments within 3 months of screening, or inability/ unwillingness to use a medically accepted contraceptive method during the study. Women who are surgically sterile or have been post-menopausal for at least 1 year will not be excluded
  * At screening, resting blood pressure (sitting or supine) lower than 90/60 or higher than 150/90, or resting heart rate lower than 45/min or higher than 100/min.
  * Imminent risk of suicidal/homicidal ideation and/or behavior with intent and/or plan.
  * Concurrent participation in a cognitive rehabilitation program, however patient will have a TBI clinician involved in directed services.
  * Subjects on a prohibited medication: monoamine oxidase inhibitors, memantine, long acting benzodiazepines (i.e., Chlordiazepoxide, Diazepam, Flurazepam)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in Severity of Depressive Symptoms | 3 weeks
  Total score on the Montgomery- Åsberg Depression Rating Scale , a semi- structured 10-item scale. Range 0-60. Higher values represent worse outcomes. The total score is obtained by summing the severity score of each item.

SECONDARY OUTCOMES:
Change in Severity of Post-traumatic Stress Disorder (PTSD) Symptoms | 3 weeks
  Total score on the PTSD Checklist for DSM-5 (PCL-5), a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. The total score is obtained by summing the score of each item.

CONTACTS AND LOCATIONS:
Locations (1):
- Minneapolis VA Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided